CLINICAL TRIAL: NCT00715741
Title: Does High Intraoperative Inspired Oxygen Reduce Postoperative Arterial Oxygen Saturation?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Harriet W. Hopf, M.D., Professor, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 29830
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Atelectasis
Keywords: atelectasis; oxygen; saturation
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Positive-Pressure Respiration; Water; Oxygen; Oxygen Saturation; Respiratory Rate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Group 1 will receive 30% oxygen plus PEEP + 3 to 5 cm Water duration of anesthesia and surgery
  Interventions: Other: FiO2 (fraction of inspired oxygen) 0.3 plus PEEP (positive end expiratory pressure) 3 -5 cm water
- 2 (Active Comparator): Group 2 will receive 30% oxygen without PEEP for the duration of anesthesia and surgery
  Interventions: Other: FiO2 0.3 without PEEP
- 3 (Active Comparator): Group 3 will receive > 90% oxygen plus PEEP + 3 to 5 cm of water for the duration of anesthesia and surgery
  Interventions: Other: FiO2 >0.9 with 3-5 cm water PEEP
- 4 (Active Comparator): Group 4 will receive > 90% oxygen and no PEEP for the duration of anesthesia and surgery
  Interventions: Other: FiO2 >0.9 without PEEP

INTERVENTIONS:
Other: FiO2 (fraction of inspired oxygen) 0.3 plus PEEP (positive end expiratory pressure) 3 -5 cm water — FiO2 (fraction of inspired oxygen) 0.3 plus PEEP (positive end expiratory pressure) 3-5 cm water
  Other Names: O2; Dioxygen; Sats; Oxygen Saturation; Pulmonary ventilation rate; Ventilation rate; Breathing rates; positive end expiratory pressure
  Arms: 1
Other: FiO2 0.3 without PEEP — FiO2 0.3 without PEEP
  Other Names: O2; Dioxygen; Sats; Oxygen Saturation; Pulmonary ventilation rate; Ventilation rate; Breathing rates
  Arms: 2
Other: FiO2 >0.9 with 3-5 cm water PEEP — FiO2 >0.9 with 3-5 cm water PEEP
  Other Names: O2; Dioxygen; Sats; Oxygen Saturation; Pulmonary ventilation rate; Ventilation rate; Breathing rates; positive end expiratory pressure
  Arms: 3
Other: FiO2 >0.9 without PEEP — FiO2 >0.9 without PEEP
  Other Names: O2; Dioxygen; Sats; Oxygen Saturation; Pulmonary ventilation rate; Ventilation rate; Breathing rates
  Arms: 4

SUMMARY:
The purpose of this study is to determine whether breathing high levels of oxygen during surgery affects oxygen levels after surgery. The second purpose of this study is to determine whether giving positive end expiratory pressure PEEP and high oxygen together affects patients oxygen levels after surgery.

DETAILED DESCRIPTION:
This is a randomized, controlled, blinded trial in patients undergoing non-abdominal surgery of the effect of intraoperative increased inspired oxygen used (FiO2>0.9 vs. FiO2 = 0.3) on non-invasive oxygen saturation (pulse oximetry, SpO2) and amount of required supplemental oxygen in the post-anesthesia care unit (PACU); arterial oxygen partial pressure (PaO2) after 45 minutes in the PACU; room air SpO2 24 hours after surgery, and amount of supplemental oxygen required 24 hours after surgery. The purpose of the study is to determine whether absorption atelectasis induced by use of inspired oxygen concentrations in excess of 90% leads to a higher risk of hypoxemia, as evidenced by room air oxygen values and the need for supplemental oxygen. The objective of this study is to determine whether high inspired oxygen (>0.8), which has been demonstrated to reduce the risk of surgical site infection in patients undergoing colon surgery and other major surgical procedures has side effects that limit its use to prevent infection in lower risk operations.

There are four groups of intraoperative ventilation management in this study. Fi02 0.3 plus PEEP, Fi02 0.3 without PEEP, Fi02 greater than 0.9 plus PEEP 3 to 5 cm of water, Fi02 greater than 0.9 without PEEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years undergoing surgery under general endotracheal anesthesia at the University of Utah Hospital Operating Room and the Huntsman Cancer Hospital Operating room who will be admitted to the hospital for at least 24 hours after surgery

Exclusion Criteria:

* Major (open) abdominal surgery
* Major spine surgery
* Craniotomy surgery
* Surgeries where electrocautery or laser devices may be used near the airway (eg tracheostomy, oral surgery) because of the risk of fire with high inspired oxygen in these cases
* Procedures planned for monitored anesthesia care (MAC) or regional without general anesthesia
* Planned airway management with a laryngeal mask airway rather than an endotracheal tube
* Procedures planned in the prone position because this increases atelectasis
* Planned postoperative intubation
* Planned postoperative care in the intensive care unit
* Recent (within 3 weeks) chemotherapy because of the increased risk of pulmonary oxygen toxicity
* History of bleomycin administration because of the increased risk of pulmonary oxygen toxicity
* Diagnosed Obstructive Sleep Apnea with home continuous pulmonary airway pressure (CPAP) use
* Home oxygen use
* Preoperative room air (RA) SpO2 <90%
* History of spontaneous pneumothorax
* Emergency surgery
* Pregnancy. Women of child-bearing age are routinely screened for pregnancy urine human chorionic gonadotropin, (HCG) on the morning of surgery. Patients with a positive result will be excluded from the study (and most likely will have their elective surgery cancelled).
* Patient refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Hopf, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Tusman G, Bohm SH, Tempra A, Melkun F, Garcia E, Turchetto E, Mulder PG, Lachmann B. Effects of recruitment maneuver on atelectasis in anesthetized children. Anesthesiology. 2003 Jan;98(1):14-22. doi: 10.1097/00000542-200301000-00006. PMID 12502973
- [Background] Belda FJ, Aguilera L, Garcia de la Asuncion J, Alberti J, Vicente R, Ferrandiz L, Rodriguez R, Company R, Sessler DI, Aguilar G, Botello SG, Orti R; Spanish Reduccion de la Tasa de Infeccion Quirurgica Group. Supplemental perioperative oxygen and the risk of surgical wound infection: a randomized controlled trial. JAMA. 2005 Oct 26;294(16):2035-42. doi: 10.1001/jama.294.16.2035. PMID 16249417
- [Background] Duggan M, Kavanagh BP. Pulmonary atelectasis: a pathogenic perioperative entity. Anesthesiology. 2005 Apr;102(4):838-54. doi: 10.1097/00000542-200504000-00021. PMID 15791115
- [Background] Myles PS, Leslie K, Chan MT, Forbes A, Paech MJ, Peyton P, Silbert BS, Pascoe E; ENIGMA Trial Group. Avoidance of nitrous oxide for patients undergoing major surgery: a randomized controlled trial. Anesthesiology. 2007 Aug;107(2):221-31. doi: 10.1097/01.anes.0000270723.30772.da. PMID 17667565

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started 06/24/2008 and ended 07/07/2009. Subjects were recruited via the Operating room schedule
Groups:
- Fi02 (Fraction of Inspired Oxygen) 0.3 With PEEP: 30% oxygen with positive end expiratory pressure (PEEP)
- Fi02 0.3 Without PEEP: 30% oxygen without PEEP
- Fi02 0.9 With PEEP: 90% oxygen plus PEEP
- Fi02 0.9 Without PEEP: 90% oxygen without PEEP
Period: Overall Study
Arm/Group | Fi02 (Fraction of Inspired Oxygen) 0.3 With PEEP | Fi02 0.3 Without PEEP | Fi02 0.9 With PEEP | Fi02 0.9 Without PEEP
Started | 25 | 25 | 25 | 25
Completed | 25 | 25 | 25 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fi02 (Fraction of Inspired Oxygen) 0.3 With PEEP | Fi02 0.3 Without PEEP | Fi02 0.9 With PEEP | Fi02 0.9 Without PEEP | Total
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 100
Age, Customized [Number; unit: participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 24 | 23 | 94
  >=65 years | 2 | 1 | 1 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (13) | 45 (12) | 46 (15) | 46 (13) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 12 | 15 | 55
  Male | 12 | 10 | 13 | 10 | 45
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 25 | 100

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Requirement to Maintain SpO2>90%
Description: Arterial oxygen saturation by pulse oximetry (SpO2) is measured while subject is lying quietly in the post anesthesia care unit (PACU) and breathing room air (RA). Oxygen is added 0.5 liters per min (LPM) at a time to maintain SpO2 >90%.
Time Frame: 45 min after emergence (tracheal extubation)
Measure: Median (Inter-Quartile Range); unit: liters per minute
Arm/Group | Fi02 (Fraction of Inspired Oxygen) 0.3 With PEEP | Fi02 0.3 Without PEEP | Fi02 0.9 With PEEP | Fi02 0.9 Without PEEP
Number analyzed (Participants) | 25 | 25 | 25 | 25
liters per minute | 1 [0.5 to 2] | 1 [0.5 to 2] | 1 [0.5 to 2] | 1 [0.5 to 2]

2. Primary Outcome: Oxygen Requirement
Description: amount of oxygen (LPM) required to maintain SpO2 >90%
Time Frame: 24 hours after tracheal extubation
Measure: Median (Inter-Quartile Range); unit: liters per min
Arm/Group | Fi02 (Fraction of Inspired Oxygen) 0.3 With PEEP | Fi02 0.3 Without PEEP | Fi02 0.9 With PEEP | Fi02 0.9 Without PEEP
Number analyzed (Participants) | 25 | 25 | 25 | 25
liters per min | 0.5 [0.5 to 2.0] | 0.5 [0.5 to 2.0] | 1.0 [0.5 to 2.0] | 0.5 [0.5 to 2.0]

3. Secondary Outcome: Arterial Oxygen Saturation by Pulse Oximetry "(SpO2)"
Description: SpO2 measured on room air or minimum supplemental oxygen to keep SpO2>90%
Time Frame: 45 min after tracheal extubation
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Fi02 (Fraction of Inspired Oxygen) 0.3 With PEEP | Fi02 0.3 Without PEEP | Fi02 0.9 With PEEP | Fi02 0.9 Without PEEP
Number analyzed (Participants) | 25 | 25 | 25 | 25
percent saturation | 95 (2) | 96 (2) | 95 (2) | 95 (2)

4. Secondary Outcome: SpO2 Postoperatively
Description: SpO2 is measured on room air or minimum oxygen required to keep SpO2>90% on the ward 24 hours after tracheal extubation.
Time Frame: 24 hours after tracheal extubation
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Fi02 (Fraction of Inspired Oxygen) 0.3 With PEEP | Fi02 0.3 Without PEEP | Fi02 0.9 With PEEP | Fi02 0.9 Without PEEP
Number analyzed (Participants) | 25 | 25 | 25 | 25
percent saturation | 95 (2) | 95 (2) | 95 (2) | 95 (2)

ADVERSE EVENTS:
Time Frame: 1 year
Description: No serious and/or non-serious adverse events were observed or assessed.
Arm/Group | Fi02 (Fraction of Inspired Oxygen) 0.3 With PEEP | Fi02 0.3 Without PEEP | Fi02 0.9 With PEEP | Fi02 0.9 Without PEEP
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
This data for this outcome measure is identical

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No